CLINICAL TRIAL: NCT06699628
Title: A Single-centre, Open-label, Phase I Trial Evaluating the Pharmacokinetics of Single Ascending Oral Doses of IRL757 in Healthy Elderly Volunteers
Brief Title: Phase I Trial Evaluating the Pharmacokinetics of Single Ascending Oral Doses of IRL757 in Healthy Elderly Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Integrative Research Laboratories AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRL757C002
Record Dates: First submitted 2024-10-22; First posted 2024-11-21 (Actual); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Not Applicable as This is a Mass Balance/Pharmacokinetic Study Performed in Healthy Subjects; Apathy
MeSH Terms: conditions — Lethargy

STUDY DESIGN:
Intervention Model Description: Ascending doses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IRL757 Dose Level 1 (Experimental): IRL757 lower dose, single dose
  Interventions: Drug: IRL757
- IRL757 Dose Level 2 (Experimental): IRL757 higher dose, single dose
  Interventions: Drug: IRL757

INTERVENTIONS:
Drug: IRL757 — IRL757 capsules

SUMMARY:
This is a phase I trial evaluating the pharmacokinetics of single ascending oral doses of IRL757 in healthy elderly volunteers.

DETAILED DESCRIPTION:
The trial is open label single oral dose trial in elderly healthy volunteers that will assess the pharmacokinetics of two dose levels of IRL757.

Eligible and consenting participants will be included in one of two dose groups, with 6 participants in each dose group.

At the screening visit, consenting subjects will be screened for eligibility according to study specific inclusion/exclusion criteria within 4 weeks before Investigational Medicinal Product (IMP) administration.

If eligible, participants will be admitted to the phase 1 clinic for the single dose administration of the IMP. All participants will receive active treatment (IRL757).

A follow-up visit will be performed for all participants, 5-10 days after IMP administration.

Blood and urine sampling will be performed for determination of pharmacokinetic parameters. Safety assessments will also be performed throughout the study: review and collection of adverse events, physical examination, suicidality ideation, electrocardiogram recording, vital signs, safety laboratory assessments.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent for participation in the trial.
* Healthy male or postmenopausal female subject at ≥ 65 and below 90 years of age.
* Weight of at least 50 kg and no more than 110 kg at screening.
* Clinically normal medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator.
* Willing to use highly effective methods of contraception

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the trial, or influence the results or the subject's ability to participate in the trial.
* GFR less than 45 mL/min at screening.
* History or present clinically significant psychiatric diagnosis, at discretion of the Investigator.
* Any suicidal ideation of type 4 or 5 in the C-SSRS in the past 3 months (i.e. active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent).
* History of seizures, including febrile seizure in childhood.
* Any clinically significant illness, medical/surgical procedure or trauma within four (4) weeks of the first administration of IMP.
* Any planned major surgery within the duration of the trial.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and Human Immunodeficiency Virus (HIV).
* After 10 minutes supine rest at the time of screening, any vital signs values outside the following ranges:

  * Systolic blood pressure above 150 mm Hg
  * Diastolic blood pressure above 90 mm Hg
  * Heart rate less than 40 or above 90 beats per minute
* Prolonged QTcF (above 450 ms for male subjects or 470 ms for female subjects), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator.
* History of severe allergy/hypersensitivity or on-going allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to IRL757.
* Use of any prescribed or non-prescribed medication including antacids, analgesics, herbal remedies, vitamins and minerals within two (2) weeks prior to the first administration of IMP
* Administration of another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical trial that included drug treatment within three (3) months of the first administration of IMP in this trial.
* Current smokers or users of nicotine products. Irregular use of nicotine (e.g. smoking, snuffing, chewing tobacco) less than three (3) times per week is allowed before screening visit.
* History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
* Positive screen for drugs of abuse at screening or on admission to the unit or positive screen for alcohol at screening or on admission to the unit prior to administration of the IMP.
* Use of anabolic steroids.
* Current excessive use of caffeine, as judged by the Investigator.
* Plasma donation within one (1) month of screening or any blood donation/blood loss more than 450 mL during the three (3) months prior to screening.
* Investigator considers the subject unlikely to comply with trial procedures, restrictions and requirements.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CTC Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- IRL757 Dose Level 1: IRL757 low dose, single dose
- IRL757 Dose Level 2: IRL757 high dose, single dose
Period: Overall Study
Arm/Group | IRL757 Dose Level 1 | IRL757 Dose Level 2
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IRL757 Dose Level 1 | IRL757 Dose Level 2 | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (4.6) | 71.2 (5.3) | 71.5 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 77.42 (13.6) | 68.2 (10.95) | 72.81 (12.72)

OUTCOME MEASURES:

1. Primary Outcome: Determination of Maximum Plasma Concentration [Cmax] of IRL757
Description: Cmax after single dosing
Time Frame: PK followed until 48 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μmol/L
Groups:
- IRL757 Dose Level 1; IRL757 Dose Level 2: IRL757, single dose
Arm/Group | IRL757 Dose Level 1 | IRL757 Dose Level 2
Number analyzed (Participants) | 6 | 6
μmol/L | 2.88 (26) | 11.42 (31)

2. Primary Outcome: Determination of the AUC of IRL757 and Its Main Metabolites
Description: AUC 0 - inf for IRL757 and main metabolites M1 and M5 determined from PK sampling 0-48h post dosing
Time Frame: PK followed until 48 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*μmol/L
Arm/Group | IRL757 Dose Level 1 | IRL757 Dose Level 2
Number analyzed (Participants) | 6 | 6
h*μmol/L
  IRL757 | 17.36 (47) | 101.3 (48)
  M1 | 1.08 (12) | 2.94 (67)
  M5 | 2.27 (42) | 10.03 (29)

3. Primary Outcome: Determination of the Time for Maximum Concentration [Tmax] of IRL757 and Its Main Metabolites
Description: Determination of the time for maximum concentration [Tmax] of IRL757 and its main metabolites M1 and M5
Time Frame: PK followed until 48 hours
Measure: Median (Full Range); unit: h
Arm/Group | IRL757 Dose Level 1 | IRL757 Dose Level 2
Number analyzed (Participants) | 6 | 6
h
  IRL757 | 0.6667 [0.333 to 1.00] | 0.75 [0.667 to 3.00]
  M1 | 0.84 [0.67 to 2.0] | 2.0 [2.0 to 4.1]
  M5 | 6.025 [5.97 to 6.03] | 6 [6 to 6]

4. Primary Outcome: Determination of the Half-life [t1/2] of IRL757 and Its Main Metabolites
Time Frame: PK followed until 48 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | IRL757 Dose Level 1 | IRL757 Dose Level 2
Number analyzed (Participants) | 6 | 6
h
  IRL757 t1/2 | 5.62 (19) | 7.44 (26)
  M1 t1/2 | 4.7 (7.7) | 6.8 (31)
  M5 IRL757 | 7.7 (29.6) | 9.95 (24.3)

5. Primary Outcome: Determination of the Renal Clearance (CLr) of IRL757
Description: Determination of the renal clearance (CLr) of IRL757 based on urine and plasma sampling over 48 h
Time Frame: PK followed until 48 hours
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | IRL757 Dose Level 1 | IRL757 Dose Level 2
Number analyzed (Participants) | 6 | 6
L/h | 0.1166 (.08364) | 0.1413 (0.09284)

6. Secondary Outcome: Evaluation of Frequency, Seriousness and Intensity of Adverse Events
Description: Total number of AEs, and total number of AEs by severity and relationship to study treatment are presented. Refer to the Adverse Events section for more information
Time Frame: From enrollment (within 4 weeks before Investigational Medicinal Product (IMP) administration, until end of follow-up (5 to 10 days after lMP administration)
Population: Total number of AEs are presented
Measure: Number; unit: AE
Groups:
- IRL757 Dose Level 2: IRL757 higher dose
Arm/Group | IRL757 Dose Level 1 | IRL757 Dose Level 2
Number analyzed (Participants) | 6 | 6
AE
  Total AEs | 1 | 3
  Treatment related AEs | 0 | 2
  Severity of AEs: MILD | 1 | 3

7. Secondary Outcome: Description of Physical Examination Findings
Description: Clinically significant abnormal findings will be summarized and categorized by dose group.
  The physical examination will include assessments of the head, eyes, ears, nose, throat, skin, thyroid, neurological, lungs, cardiovascular, abdomen (liver and spleen), lymph nodes and extremities.
Time Frame: Until 5-10 days after IMP administration
Measure: Number; unit: Clinically significant abnormalities
Arm/Group | IRL757 Dose Level 1 | IRL757 Dose Level 2
Number analyzed (Participants) | 6 | 6
Clinically significant abnormalities
  Abnormal Clinically Significant findings | 0 | 0

8. Secondary Outcome: Description of Electrocardiogram Findings
Description: Following parameters will be measured/calculated: heart rate, PR, QRS, QT and QTc intervals. The measures will be described as "normal", "abnormal, not clinically significant", or "abnormal, clinically significant". These will be summarized and categorized by dose group.
Time Frame: Until 5-10 days after IMP administration
Measure: Count of Participants; unit: Participants
Arm/Group | IRL757 Dose Level 1 | IRL757 Dose Level 2
Number analyzed (Participants) | 6 | 6
Participants
  Abnormal, not clinically significant | 1 | 1
  Abnormal, clinically significant | 0 | 0

9. Secondary Outcome: Description of Vital Signs Findings
Description: The following parameters will be measured as vital signs: systolic and diastolic blood pressure, heart rate and respiratory rate. Clinically significant findings will be summarized by dose group.
Time Frame: Until 5-10 days after IMP administration
Measure: Number; unit: Clinically significant changes
Arm/Group | IRL757 Dose Level 1 | IRL757 Dose Level 2
Number analyzed (Participants) | 6 | 6
Clinically significant changes | 0 | 0

10. Secondary Outcome: Description of Safety Laboratory Measurements
Description: Common laboratory parameters will be assessed: clinical biochemistry panel (including for example, ALAT, ASAT, ALP, CRP, CK, Calcium, Potassium, Sodium,...), hematology panel (including white blood cell differential count), coagulation parameters (INR, APTT).
  Safety laboratory data will be summarized by dose group. Safety laboratory interpretations (abnormal, significant) will be summarized by dose groups, using frequency tables.
Time Frame: Until 5-10 days after IMP administration
Measure: Number; unit: Clinically significant abnormalities
Arm/Group | IRL757 Dose Level 1 | IRL757 Dose Level 2
Number analyzed (Participants) | 6 | 6
Clinically significant abnormalities | 0 | 0

11. Secondary Outcome: Description of C-SSRS (Columbia Suicide Severity Rating Scale) Findings
Description: A physician rates an individual's degree of suicidal ideation on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent". Any abnormal finding will be listed.
Time Frame: Until 5-10 days after IMP administration
Measure: Number; unit: Abnormal findings
Arm/Group | IRL757 Dose Level 1 | IRL757 Dose Level 2
Number analyzed (Participants) | 6 | 6
Abnormal findings | 0 | 0

ADVERSE EVENTS:
Time Frame: From enrollment (within 4 weeks before Investigational Medicinal Product (IMP) administration, until end of follow-up (5 to 10 days after lMP administration)
Arm/Group | IRL757 Dose Level 1 | IRL757 Dose Level 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IRL757 Dose Level 1 (N=6) | IRL757 Dose Level 2 (N=6)
Headache (Nervous system disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-10-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT06699628/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT06699628/SAP_001.pdf